CLINICAL TRIAL: NCT00393094
Title: A Phase II Trial of Bevacizumab and Irinotecan for Patients With Recurrent High-Grade Gliomas Immediately Following Tumor Progression After Treatment w/Bevacizumab Alone: A Companion Trial to NCI Study 06-C-0064 (NCT00271609)(Bevacizumab Alone for Recurrent Gliomas)
Brief Title: Bevacizumab and Irinotecan to Treat Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to the limitations of accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Howard A. Fine, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060250; 06-C-0250
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: High-Grade Gliomas
Keywords: Brain Tumor; Chemotherapy; Progression; Radiotherapy; Antiangiogenesis; Glioma
MeSH Terms: conditions — Brain Neoplasms; Disease Progression; Glioma | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab & Irinotecan Patients (Experimental): Bevacizumab - 10 mg/kg intravenous injection Irinotecan - 125 mg/m^2 if patient is on a non-enzyme inducing anti-epileptic drugs 340 mg/m^2 if patient is on enzyme inducing anti-epileptic drugs every two weeks on a 4 week cycle
  Interventions: Biological: Bevacizumab; Drug: Irinotecan hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — 10 mg/kg intravenous injection
  Other Names: rhuMAb VEGF
Drug: Irinotecan hydrochloride — 125 mg/m^2 if patient is on a non-enzyme inducing anti-epileptic drugs 340 mg/m^2 if patient is on enzyme inducing anti-epileptic drugs every two weeks on a 4 week cycle
  Other Names: irinotecan hydrochloride trihydrate; CPT-11; Camptosar

SUMMARY:
Background:

* Bevacizumab is a genetically engineered antibody that blocks the growth of new blood vessels in tumors. It has shown activity against human brain tumors in laboratory tests and human clinical trials.
* Irinotecan causes damage to the deoxyribonucleic acid (DNA) in cancer cells so that the cells cannot reproduce or repair themselves. It is approved for treating patients with colorectal cancer.
* Bevacizumab and irinotecan in combination are more effective against colon cancer than either drug alone.

Objectives:

* To determine the safety of bevacizumab and irinotecan and any side effects associated with the combination of the two drugs when given to patients with high grade gliomas.
* To determine if the combination of bevacizumab and irinotecan can help patients with brain tumors that have grown after treatment with bevacizumab alone.

Eligibility:

-Patients 18 years of age and older who have been treated on National Cancer Institute (NCI) trial 06-C-0064 (NCT00271609), "Bevacizumab Alone for Recurrent Gliomas," and whose tumor has progressed.

Design:

Participants receive infusions of bevacizumab and irinotecan through a vein once every 2 weeks in 4-week treatment cycles, plus the following procedures:

* History, physical and neurological examinations every 2 weeks for the first treatment cycle and then every 4 weeks
* Magnetic Resonance Imaging (MRI) scan of the head every 4 weeks.
* Routine lab every week.
* Quality-of-life questionnaire every 4 weeks

DETAILED DESCRIPTION:
Background:

* Bevacizumab is a humanized IgG1 monoclonal antibody (MAb) that binds all biologically active isoforms of human vascular endothelial growth factor (VEGF, or VEGF-A) with high affinity (kd = 1.1 nM ). The antibody consists of a human IgG1 framework and the antigen-binding complementarity-determining regions from the murine anti-VEGF MAb A.4.6.1.
* Irinotecan is a semisynthetic derivative of camptothecin that possesses greater aqueous solubility, greater in vitro and in vivo activity, and is associated with less severe and more predictable toxicity than camptothecin.
* We now propose treating patients whose tumors progress on our bevacizumab alone protocol with the combination of bevacizumab with irinotecan. We believe that this trial design has significant power to detect a true synergistic effect between the two agents given that the single agent activity of irinotecan is so low in patients with recurrent malignant gliomas (2-5% response rate) and the patients being treated on this trial will have tumors that have already progressed through bevacizumab.

Objective:

* To establish data and safety regarding the anti-tumor activity of bevacizumab plus irinotecan in patients with recurrent high-grade gliomas that have progressed on bevacizumab alone as determined by objective radiographic response rate.
* To determine the 6 month progression-free survival of treated patients and to characterize the pattern of changes in the number of endothelial progenitor cells over time and across patients.
* To obtain preliminary data regarding how response to treatment (stable disease or radiographic response) effects monthly measurements of quality of life while on study.

Eligibility:

* Patients must have been treated on the National Cancer Institute (NCI) trial 06-C-0064; bevacizumab alone for recurrent gliomas and now have evidence for tumor progression by magnetic resonance imaging (MRI) scan.
* Patients with histologically proven intracranial malignant glioma.

Design:

-Patients will be treated with bevacizumab by intravenous injection at a dose of 10mg/kg and irinotecan at a dose of 125 mg/m^2 for patients on non-enzyme-inducing anti-epileptic drugs (NEIAED) and 340 mg/m^2 for patients on enzyme-inducing anti-epileptic drugs (EIAED) every two weeks on a 4-week cycle.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have been treated on the National Cancer Institute (NCI) trial 06-C-0064 (NCT00271609); bevacizumab alone for recurrent gliomas and now have evidence for tumor progression by magnetic resonance imaging (MRI) scan.

Patients with histologically proven intracranial malignant glioma will be eligible for this protocol. Malignant glioma include glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).

Patients must have evidence for tumor progression by MRI or computed tomography (CT) scan. This scan should be performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline magnetic resonance (MR)/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.

All patients or their previously designated durable power of attorney (DPA) (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.

Patients must have a Karnofsky performance status of greater than or equal to 60.

Patients must not be more than 4 weeks since their last bevacizumab treatment and may have received no form of treatment (i.e. radiation, chemotherapy, surgery, investigational therapy) for their progressive tumor between their last bevacizumab treatment and enrollment of this companion trial.

Patients must have adequate bone marrow function (white blood cell (WBC) greater than or equal 3,000/microl, absolute neutrophil count (ANC) greater than or equal to1,500/mm^3, platelet count of greater than to or equal 100,000/mm^3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (serum glutamic oxaloacetic transaminase (SGOT) and bilirubin less than 2.5 times upper limits of normal (ULN)), and adequate renal function (creatinine less than 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy.

This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race.

Urine protein should be screened by dipstick or urine analysis for Urine Protein Creatinine (UPC) ratio. For proteinuria greater than or equal to 1+ or urine protein:creatinine UPC ratio greater than 1.0, 24-hour urine protein should be obtained and the level should be less than 1000 mg for patient enrollment.

Subjects must be willing and able to practice adequate contraception.

EXCLUSION CRITERIA:

Concurrent use of other standard chemotherapeutics or investigative agents.

Patients who have an active infection.

Pregnant (positive pregnancy test) or nursing women. Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy.

Concurrent anti-coagulation or anti-platelet medication (including aspirin, non-steroidal anti-inflammatories, cyclooxygenase-2 (COX-2) inhibitors).

Serious or non-healing wound, ulcer or bone fracture.

History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.

Invasive procedures defined as follows:

* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to day (D)1 therapy

Patients with clinically significant cardiovascular disease:

* History of cerebrovascular accident (CVA) within 6 months
* Uncontrolled hypertension (greater than 150/100 mmHg)
* Myocardial infarction or unstable angina within 6 months
* New York heart association grade II or greater congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Unstable angina pectoris
* Clinically significant peripheral vascular disease

Clinical evidence of bleeding diathesis or coagulopathy.

Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Fine, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker D, Wright E, Nguyen K, Cannon L, Fain P, Goldgar D, Bishop DT, Carey J, Baty B, Kivlin J, et al. Gene for von Recklinghausen neurofibromatosis is in the pericentromeric region of chromosome 17. Science. 1987 May 29;236(4805):1100-2. doi: 10.1126/science.3107130.
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991
- [Background] Kreisl TN, Kim L, Moore K, Duic P, Royce C, Stroud I, Garren N, Mackey M, Butman JA, Camphausen K, Park J, Albert PS, Fine HA. Phase II trial of single-agent bevacizumab followed by bevacizumab plus irinotecan at tumor progression in recurrent glioblastoma. J Clin Oncol. 2009 Feb 10;27(5):740-5. doi: 10.1200/JCO.2008.16.3055. Epub 2008 Dec 29. PMID 19114704
- [Result] Kreisl TN, Zhang W, Odia Y, Shih JH, Butman JA, Hammoud D, Iwamoto FM, Sul J, Fine HA. A phase II trial of single-agent bevacizumab in patients with recurrent anaplastic glioma. Neuro Oncol. 2011 Oct;13(10):1143-50. doi: 10.1093/neuonc/nor091. Epub 2011 Aug 24. PMID 21865400
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0250.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Period: Period1Bevacizumab & Irinotecan Patients
Arm/Group | Enrollment Until Prior to Treatment
Started | 31
Completed | 30
Not Completed | 1
Not completed — Disease progression before treatment | 1
Period: Disease Progression After Trtmt: Onstudy
Arm/Group | Enrollment Until Prior to Treatment
Started | 30
Completed | 29
Not Completed | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrollment Until Prior to Treatment
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 46.96 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rate (Malignant Glioma Participants)
Description: Definition of response: complete response (CR) is the complete disappearance of all measurable and evaluable disease. Partial response (PR) is greater than or equal to a 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions. Stable/No response (SD, NR)does not qualify for CR, PR, or progression. Progression is a 25% increase in the sum of products of all measurable lesions (or two target lesions if too numerous over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline.
Time Frame: 23 months (date of first enrollment to 1 month after last progression)
Population: Analysis is per protocol (N=30), excluding the 1 patient who progressed and withdrew consent prior to any treatment but after enrollment.
Measure: Number; unit: Percent of participants
Arm/Group | Enrollment Until Prior to Treatment
Number analyzed (Participants) | 30
Percent of participants
  Partial response | 0
  Complete response | 0
  Stable disease | 16.7
  Progressive disease | 83.3

2. Primary Outcome: Number of Participants With Toxicity as Measured by The National Cancer Institute (NCI) Common Toxicity Criteria v. 3.0.
Description: Here is the number of participants with any toxicity, defined as any adverse events possibly, probably or definitely related to the investigational drugs. For the detailed list of investigational new drug (IND)-related toxicities and other serious adverse events, see the adverse event module.
Time Frame: 23 months (date of first enrollment to 1 month after last progression)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Enrollment Until Prior to Treatment
Number analyzed (Participants) | 30
Participants | 27

3. Primary Outcome: Radiographic Response Rate (Anaplastic Glioma Participants)
Description: as for outcome 1
Time Frame: 23 months (date of first enrollment to 1 month after last progression)
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Groups:
- Bevacizumab & Irinotecan Anaplastic Glioma Pts: Enrollment: Bevacizumab - 10 mg/kg intravenous injection Irinotecan - 125 mg/m^2 if patient is on a non-enzyme inducing anti-epileptic drugs 340 mg/m^2 if patient is on enzyme inducing anti-epileptic drugs every two weeks on a 4 week cycle Anaplastic gliomas are classified by the World Health Organization (WHO) as grade 3 malignant tumors and include the anaplastic astrocytoma, anaplastic oligodendroglioma, and anaplastic oligoastrocytoma or mixed glioma.
Arm/Group | Bevacizumab & Irinotecan Anaplastic Glioma Pts: Enrollment
Number analyzed (Participants) | 30
Percent of participants
  Partial response | 0
  Complete response | 0
  Stable disease | 30
  Progressive disease | 70

4. Primary Outcome: Radiographic Response Rate (Glioblastoma Multiforme Participants)
Description: as for outcome 1
Time Frame: 23 months (date of first enrollment to 1 month after last progression)
Measure: Number; unit: Percent of participants
Groups:
- Bevacizumab & Irinotecan Glioblastoma Multiforme: Enrollment: Bevacizumab - 10 mg/kg intravenous injection Irinotecan - 125 mg/m^2 if patient is on a non-enzyme inducing anti-epileptic drugs 340 mg/m^2 if patient is on enzyme inducing anti-epileptic drugs every two weeks on a 4 week cycle Glioblastoma multiforme- is a fast growing type of central nervous system tumor that forms from glial (supportive) tissue of the brain and spinal cord and has cells that look very different from normal cells. Glioblastoma multiforme usually occurs in adults and affects the brain more often than the spinal cord. Also called GBM, glioblastoma, and grade IV astrocytoma.
Arm/Group | Bevacizumab & Irinotecan Glioblastoma Multiforme: Enrollment
Number analyzed (Participants) | 20
Percent of participants
  Partial response | 0
  Complete response | 0
  Stable disease | 10
  Progressive disease | 90

ADVERSE EVENTS:
Time Frame: 23 months
Arm/Group | Enrollment Until Prior to Treatment
Serious Adverse Events (participants affected / at risk) | 9/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Until Prior to Treatment (N=30)
Death not associated with CTCAE term: Death Progression NOS (General disorders) | 1 (1)
Hemoglobin (Investigations) | 2 (2)
Neurology: Seizure (Nervous system disorders) | 5 (5)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Leukocytes (total white blood count (WBC)) (Blood and lymphatic system disorders) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2)
Neutrophils/granulocytes (absolute neutrophil count (ANC)/absolute granulocyte count (AGC)) (Blood and lymphatic system disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) (Metabolism and nutrition disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Until Prior to Treatment (N=30)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 5 (6)
Alkaline phosphatase (Investigations) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 18 (22)
Hemoglobin (Investigations) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 9 (12)
Lymphopenia (Investigations) | 1 (3)
Nausea (Gastrointestinal disorders) | 10 (13)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 (13)
Pain: head/headache (Nervous system disorders) | 3 (3)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (12)
Platelets (Investigations) | 5 (9)
Vomiting (Gastrointestinal disorders) | 5 (5)
Cytokine release syndrome/acute infusion reaction (General disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hemorrhage, central nervous system (CNS) (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, genitourinary (GU) retroperitoneum (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: Nose (Blood and lymphatic system disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Evaluating combination therapy, 19 GBM patients were enrolled. Accrual was terminated after it became clear that we could not reach our efficacy rule of 3 or more of 29 patients responding. The AG arm never fully accrued before the study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No